CLINICAL TRIAL: NCT04893382
Title: Deciphering the Inflammatory Consequences of Crystalloids Used in the Resuscitation of Severely Burned Patients
Brief Title: Inflammatory Consequences of Crystalloids in Severely Burned Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funds and participants
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20.443
Record Dates: First submitted 2021-05-12; First posted 2021-05-19 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Burns
Keywords: Resuscitation; Crystalloids; Inflammation
MeSH Terms: conditions — Burns; Inflammation | interventions — Plasmalyte A; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Patients admitted to the severely burned unit will be randomized by the research nurse to either received PlasmaLyte or Ringer's Lactate. Research Nurse will then advise the treating team.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PlasmaLyte (Experimental): Seven (7) severely burned patients will be infused with PlasmaLyte (following randomization) during the resuscitation period following admission to the ICU. 50mL of blood will be withdrawn before the first infusion and for the following days (Day 1-2-5 and 10) in order to isolate neutrophils and monocytes. Plasma will be preserved for future cytokines characterization.
  Interventions: Procedure: PlasmaLyte for fluid resuscitation
- Ringer's Lactate (Experimental): Seven (7) severely burned patients will be infused with Ringer's Lactate (following randomization) during the resuscitation period following admission to the ICU. 50mL of blood will be withdrawn before the first infusion and for the following days (Day 1-2-5 and 10) in order to isolate neutrophils and monocytes. Plasma will be preserved for future cytokines characterization.
  Interventions: Procedure: Ringer's Lactate for fluid resuscitation

INTERVENTIONS:
Procedure: PlasmaLyte for fluid resuscitation — Fluid resuscitation is a critical and essential part in the treatment of severely burned patients. Patients randomized for this arm will be submitted to PlasmaLyte infusion (as clinically prescribed).
  Arms: PlasmaLyte
Procedure: Ringer's Lactate for fluid resuscitation — Fluid resuscitation is a critical and essential part in the treatment of severely burned patients. Patients randomized for this arm will be submitted to Ringer's Lactate infusion (as clinically prescribed).
  Arms: Ringer's Lactate

SUMMARY:
This is a pilot study, but the investigators will also observe key immunological events with potential significance. The global objective is to study the inflammatory profiles of PlasmaLyte and Ringer's Lactate used in the initial massive fluid resuscitation of severely burned patients. On the long term, the investigators will identify the crystalloid that prevents hyperactivation of macrophages and death of severely burned patients.

DETAILED DESCRIPTION:
The investigators have 4 specific objectives. First, the investigators will compare the activation profiles of macrophages and neutrophils in patients admitted to the severely burned unit with regards to the crystalloids used. Secondly, the investigators will assess the differences in the SOFA scores according to the crystalloids used. Thirdly, the investigators will evaluate the impact of crystalloids in the quality of skin grafts performed on severely burned patients. Lastly, with the help of a patient partner, the investigators will determine the right immunological terminology of the study for a non-scientific population.

ELIGIBILITY:
Inclusion Criteria:

* admission to the CHUM
* more than 20% of burned area
* first blood withdrawal in the first 24 hours following burn

Exclusion Criteria:

* immunosuppression
* chemotherapy 6 months before admission
* radiotherapy 6 months before admission
* autoimmune diseases
* neoplasia
* pregnancy
* severe infections
* cardiac dysfunctions
* renal dysfunction
* hepatic dysfunctions
* Hepatitis C
* HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-10-17 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Change in monocyte phenotype from admission to day 10 | Pre-infusion to day 10 post-infusion
  Following blood draws, monocytes will be subjected to flow cytometry for phenotype evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Cailhier, MD, Principal Investigator — CRCHUM
Locations (1):
- CHUM, Montreal, Quebec, Canada